CLINICAL TRIAL: NCT07046091
Title: Effects of a 20-Minute Mindfulness-Based Breathing Exercise on Dyspnea, Fatigue, and Sleep Quality in Patients With Heart Failure
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Gui Dural, Associate professor, Firat University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FUGDRL-001
Record Dates: First submitted 2025-02-07; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-02

CONDITIONS: Heart Failure; Heart Failure - NYHA II - IV
Keywords: heart failure; mindfulness; dsypnea; fatigue; sleep quality
MeSH Terms: conditions — Heart Failure; Fatigue; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention phase (Experimental): Mindfulness-based approaches help to focus attention and teach individuals strategies for coping with challenging situations, accepting experiences, building self-confidence, and disengaging. Mindfulness-based practices increase an individual's level of awareness and distance them from current or potential stress factors. In recent years, non-pharmacological complementary and integrative interventions have become more widely used in disease management. Studies supporting the use of mindfulness-based interventions, particularly for the management of acute and chronic pain, have demonstrated biological and psychological improvements. In this study, the aim of the 20-minute mindfulness-based breathing exercise program is to reduce dyspnea and fatigue levels and improve sleep quality in heart failure patients who face many challenging situations. After a pre-test, the experimental group will receive the mindfulness-based breathing exercise program. The program will last for 6 weeks, with
  Interventions: Behavioral: 20-minute mindfulness-based breathing exercise
- control phase (Experimental): No intervention would be applied to patients in this group and only pre-test and post-test data would be collected.
  Interventions: Behavioral: Control (Standard treatment)

INTERVENTIONS:
Behavioral: 20-minute mindfulness-based breathing exercise — Mindfulness-based approaches help to focus attention and teach individuals strategies for coping with challenging situations, accepting experiences, building self-confidence, and disengaging. Mindfulness-based practices increase an individual's level of awareness and distance them from current or potential stress factors. In recent years, non-pharmacological complementary and integrative interventions have become more widely used in disease management. Studies supporting the use of mindfulness-based interventions, particularly for the management of acute and chronic pain, have demonstrated biological and psychological improvements. In this study, the aim of the 20-minute mindfulness-based breathing exercise program is to reduce dyspnea and fatigue levels and improve sleep quality in heart failure patients who face many challenging situations. After a pre-test, the experimental group will receive the mindfulness-based breathing exercise program. The program will last for 6 weeks, with e
  Arms: Intervention phase
Behavioral: Control (Standard treatment) — No intervention would be applied to patients in this group and only pre-test and post-test data would be collected.
  Arms: control phase

SUMMARY:
Heart failure (HF) is a chronic condition that leads to incapacity. Despite significant progress in optimizing pharmacological treatment for HF patients, the personal and social burden of this disease is still characterized by debilitating symptoms and rehospitalizations. Today, many patients with heart failure use non-pharmacological methods for managing common symptoms. Due to the increased interest in non-pharmacological methods among individuals in society, it has become essential for healthcare professionals, including nurses as part of the healthcare team, to play a role in these methods to meet the health needs of the community.

One of the interventions nurses can offer for symptom management is mindfulness-based breathing exercises. In this mind-body-based practice, attention is focused on the breath, helping individuals develop awareness of their negative thoughts and emotions.

The study population will consist of patients admitted to the Cardiology Department of Firat University Hospital. The sample size was determined by a power analysis, with a 0.05 margin of error, a 0.95 confidence interval, and a 0.5 effect size, representing 80% of the population, resulting in 72 patients for both the experimental and control groups. Data collection tools for the study will include a Personal Information Form, the Dyspnea-12 Scale, the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Scale, and the Richard-Campbell Sleep Scale. SPSS (Statistical Programme for Social Sciences) software will be used to analyze the data obtained from the study.

The aim of this study is to determine the effects of a 20-minute mindfulness-based breathing exercise on dyspnea, fatigue, and sleep quality in patients with heart failure.

DETAILED DESCRIPTION:
Heart failure, with a global prevalence of 26 million, is a leading cause of morbidity and mortality. Compared to its corrected incidence, the prevalence of heart failure is expected to rise due to the aging population. Hospital admissions due to heart failure impose a significant socioeconomic burden, especially due to increasing healthcare costs. It is estimated that more than half of the total expenditures related to heart failure are due to hospital admissions, while pharmacotherapy contributes to 18% of the cost.

Heart failure (HF) is a chronic condition that leads to incapacity. Despite significant progress in optimizing pharmacological treatment for HF patients, the personal and social burden of this disease remains characterized by debilitating symptoms and rehospitalizations. Generalized muscle atrophy, including inspiratory muscle atrophy, is often observed in patients with heart failure. Weakness of the respiratory muscles during exercise and activity can lead to fatigue and shortness of breath.

Dyspnea, early fatigue, exercise intolerance, and reduced life expectancy are common symptoms and signs of heart failure, characterized by the inability of the heart to meet the metabolic demands of tissues. In a study conducted on patients with heart failure, the frequency of severe dyspnea was reported as 69%. The mechanism of dyspnea is multifactorial. Dyspnea can exacerbate fatigue by limiting daily activities in HF patients .

Fatigue is also a prototypical symptom of heart failure. In a study, 59% of HF patients reported moderate to severe fatigue. Fatigue is a reflection of muscle hypoperfusion and is an indicator of reduced cardiac output, with its intensity related to depression, muscle dysfunction, and symptoms of anemia. Fatigue is also an independent predictor of increased cardiac readmission and mortality rates in HF patients. It can be explained by clinical factors such as age, anemia, poor sleep quality, reduced exercise capacity, dyspnea, and psychosocial distress.

Changes in sleep patterns in heart failure patients can negatively affect the prognosis of the disease. Pharmacological methods are the most known and frequently used treatments for patients with sleep problems. However, it is also known that long-term use of medications for sleep problems has the potential to cause serious side effects. Therefore, in recent years, non-pharmacological methods are also being utilized to improve sleep quality in individuals with sleep issues.

Non-pharmacological treatments can be beneficial for HF patients. Research evidence shows that non-pharmacological interventions, especially breathing training, have benefits on dyspnea and anxiety in patients with heart failure. For example, a mindfulness-based psychoeducation intervention, which focuses on cognitively separating bodily sensations from stimulated thoughts and emotions, has been shown to significantly reduce anxiety in patients with chronic heart failure and improve their symptoms. Mindfulness involves consciously paying attention to the present moment in a non-reactive way. It has been shown to reduce stress, anxiety, and depression while improving sleep. Although there is growing evidence supporting the application of mindfulness in various chronic diseases, its benefit in reducing dyspnea remains uncertain. However, most of the evidence on the benefits of mindfulness comes from traditional 6-8 week mindfulness programs. Short mindfulness practices, lasting 5-30 minutes, warrant further research. Recent studies have shown that a single 20-minute mindful breathing session significantly reduced dyspnea in patients with chronic lung disease and decompensated heart failure.

Mindful breathing is an exercise that involves paying attention to one's breath without distraction from external or internal experiences. This maneuver has been shown to relieve distress in patients in palliative care and reduce dyspnea in patients with chronic lung disease. A recent study reported that an 8-week mindfulness-based intervention reduced dyspnea, fatigue, and dizziness symptoms in symptomatic congestive heart failure outpatients compared to traditional treatment alone.

Short mindfulness practices require less energy and time from patients and have the potential to create more sustainable habits when practiced regularly. However, evidence for their effectiveness in reducing fatigue is still lacking. A literature review found that there is insufficient research on mindfulness-based breathing exercises for heart failure patients. This study is expected to contribute to the nursing literature. The aim of this study is to determine the effects of a 20-minute mindfulness-based breathing exercise on dyspnea, fatigue, and sleep quality in patients with heart failure.

ELIGIBILITY:
Inclusion Criteria

* Over 18 years of age
* Able to communicate effectively
* No psychiatric disorders Exclusion Criteria
* Patients with communication problems
* Patients with psychiatric disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
dyspnea severity | Baseline and 6 weeks after intervention
  Dyspnea Severity Measurement Tool: Dyspnea-12 Scale Time Frame: [Measurement time, e.g., "After a 20-minute mindfulness-based breathing exercise"] Unit of Measure: [Unit of measure, e.g., "scores"] Scale Title: Dyspnea-12 Scale Scale Range: [0] - [12] Interpretation: Higher scores indicate worse outcomes.
Fatigue Severity | Baseline and 6 weeks after intervention
  Fatigue Measurement Tool: FACIT-F Scale Time Frame: [Measurement time, e.g., "After mindfulness-based breathing exercise intervention"] Unit of Measure: [Unit of measure, e.g., "scores''] Scale Title: FACIT-F Scale (Functional Assessment of Chronic Illness Therapy - Fatigue) Scale Range: [0] - [52] Interpretation: Higher scores indicate higher levels of fatigue.
Sleep quality | Baseline and 6 weeks after intervention
  Sleep Quality Measurement Tool: Richard-Campbell Sleep Scale Time Frame: [Measurement time, e.g., "After mindfulness-based breathing exercise"] Unit of Measure: [Unit of measure, e.g., "scores"] Scale Title: Richard-Campbell Sleep Scale Scale Range: [0] - [21] Interpretation: Higher scores indicate better outcomes.

IPD SHARING:
Plan to Share IPD: Undecided